CLINICAL TRIAL: NCT07311486
Title: BLOOD BIOMARKERS TO IMPROVE MANAGEMENT OF MILD TRAUMATIC BRAIN INJURY IMPLIMENTACIÓN STUDY
Brief Title: Implementation of Biomarker-Based Care for mTBI - IMPACTS-BRAINI Study
Acronym: IMPACTS-BRAINI
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Alfonso Lagares Gómez-Abascal, Professor of Neurosurgery, Head of Department Neurosurgery, Hospital Universitario 12 de Octubre
Other Study IDs: TP25/0144
Record Dates: First submitted 2025-12-08; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Mild Traumatic Brain Injury (mTBI)
Keywords: Biomarker; GFAP; UCH-L1; Implementation
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implemetation Mild TBI cohort: Mild TBI patients managed before the implementation of the combined GFAP UCH-L1 test
- Post-implementation Mild TBI cohort: Prospective Mild TBI patients managed following a clinical pathway including the use of the combined GFAP UCH-L1 diagnostic test in a real world enviroment
  Interventions: Diagnostic Test: GFAP and UCH-L1

INTERVENTIONS:
Diagnostic Test: GFAP and UCH-L1 — Serum test to measure the concentration of GFAP and UCH-L1
  Groups: Post-implementation Mild TBI cohort

SUMMARY:
This study aims to evaluate the real-world applicability and clinical added value of a new management pathway for patients presenting to the emergency department (ER) with mild traumatic brain injury (mTBI). The pathway includes the use of the VIDAS® TBI in vitro diagnostic assay, which measures the blood biomarkers GFAP and UCH-L1 within 12 hours of injury to determine whether a CT scan is necessary.

The study seeks to answer two primary questions:

1. Safety and effectiveness: Whether the VIDAS® TBI test can safely and accurately rule out the need for head CT in mTBI patients in routine emergency care.
2. Clinical and operational impact: Whether incorporating this test reduces the number of CT scans performed and shortens ER length of stay for patients with mild TBI.

To assess these outcomes, researchers will compare patient management using the new biomarker-based pathway to a historical cohort of mTBI patients who were managed without the biomarker test.

DETAILED DESCRIPTION:
GENERAL OBJECTIVE To assess the applicability and added value of a new clinical management pathway for patients with mild TBI presenting to the emergency department (ER), including the use of an in vitro diagnostic assay measuring the biomarkers GFAP and UCH-L1 in the serum, within the first 12 hours post-injury, to rule out the need for CT scan in mild TBI patients.

PRINCIPAL OBJECTIVE To evaluate the diagnostic performance of the VIDAS TBI (GFAP&UCH-L1) test in determining the need for CT-scan in patients with mild TBI admitted to the ER of Hospital 12 de Octubre.

To determine the safety of a management protocol including the use of the VIDAS GFAP&UCH-L1 test for patients with mTBI, in terms of complications or unforeseen neurological deterioration following the injury.

To estimate the reduction of CTs achieved using the biomarker test, by comparison with the management of TBI during the six months preceding the study (reference pathway).

METHODOLOGY The study will compare the different outcome measures between a historic group obtained 6 months before the initiation of the new management protocol and the group of patients admitted in the ER with a diagnosis of a mTBI after the initiation of the new bundle of care. Therefore the methodology of the study is an ambispective (or mixed) cohort study with historical controls.

The combined GFAP&UCH-L1 test has been included in the new bundle of care of mTBI for the management in the ER of all patients with mTBI. In summary the test will be performed to all patients with mTBI admitted to the ER of Hospital 12 de Octubre and included in the new management pathway of patients with mTBI incorporated in our hospital. All patients suffering a mTBI(GCS 15-13) and admitted within 12 hours of the TBI will be included in this pathway. If the patient is included in this pathway, the prescription of cranial CT will be performed following the results of the VIDAS TBI test if the patient has had a significant TBI and a GCS of 14 or 15. Those patients with GCS of 13 or a focal neurological deficit will receive both biomarkers and CT for their management during the study period. The VIDAS TBI test interpretation as defined by the manufacturer, bioMérieux, takes into account the responses of the two biomarkers: the VIDAS TBI test is negative if the two markers GFAP and UCH-L1 are negative (below the previously defined threshold concentration for each of the biomarkers). The test is positive if at least one of the two GFAP or UCH-L1 biomarkers is positive (beyond the threshold concentration). This test is already CE marked and has already been tested on a large number of European patients and has demonstrated good safety and reliability profiles.

STUDY POPULATION Mild TBI patients with significant brain trauma admitted in the ER of Hospital 12 de Octubre

NUMBER OF SUBJECTS The implementation study will last for 6 months. The number of patients that are normally treated for this pathology is around 3000 patients each year. During the 6 months of the study around 1000 patients will at least be triaged for mild TBI EXPECTED IMPACT This study will demonstrate the feasibility of using a bundle of care based on the determination of blood-based brain biomarkers in the management of patients with mTBI, in a real-life setting. It will also determine the time needed for obtaining results of these blood derived biomarkers and if there is reduction in associated cost and CT prescription related to its use related to a historical control cohort.

ELIGIBILITY:
Inclusion Criteria:

* -All adult patients suffering mild TBI:( Defined by at least criterion a) and d) and one or more of the other criteria)

  1. The presence of a plausible traumatic mechanism observed/or related by the patient´s recount of the injury event.
  2. Presence of one or more clinical signs attributable to brain injury: Loss of consciousness immediately following injury, alteration of mental status immediately following the injury, posttraumatic amnesia or any neurological abnormality.
  3. At least two acute symptoms related to the injury: feeling confused or disoriented, headache, nausea, vomiting, dizziness, vision problems, memory problems, emotional lability or irritability.
  4. a GCS between 15 and 13, at least 30 minutes after injury.
* Blood sample obtained ≤12 h after injury and ideally before any imaging prescription.

Exclusion Criteria:

* · GCS 3-12 on admission

  * Age Below 18 years
  * Time of injury unknown
  * Time to injury exceeding 12 hours
  * Primary admission for non-traumatic neurological disorder (e.g., stroke, spontaneous, intracranial hematoma)
  * Penetrating head trauma
  * Patient with mechanical ventilation from the trauma scene or prehospital management
  * Venipuncture not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild traumatic brain injured patients admitted in the ER less than 12 hours after injury
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the biomarker test | 12 hours after mild TBI
  Sensitivity, specificity and NPV of the combined biomarker test to determine the presence of lesions on CT
Proportion (%) of CT scan prescribed in the ER over the period of the study for patients with mTBI | 12 hours after mild TBI
  Proportion of patients in whom a CT scan has been performed for screening of intracranial lesiones

SECONDARY OUTCOMES:
Time spent in the ED | 12 hours after mild TBI
  Time from admission to discharge. Time from admission to sample obtention. Time from venipuncture to availability of biomarker results.
Compliance with proposed algorithm | 12 hours after mild TBI
  Number of patients in whom a CT scan has been performed despinte negative biomarker test

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Lagares, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (de-identified) that underlie the results reported in this study will be made available only upon request, after publication of the main results, to researchers who provide a methodologically sound proposal. Data will be shared in accordance with applicable ethical and regulatory requirements, and a data-sharing agreement will be required.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data will be available from 6 months to 5 years after publication of the study results, upon reasonable request. After this period, data availability cannot be guaranteed.
Access Criteria: Access to de-identified individual participant data will be granted only upon reasonable request to researchers who submit a methodologically sound proposal and whose intended use is consistent with the study objectives and ethical standards. Requestors must sign a data-sharing agreement outlining conditions for data use, confidentiality, and prohibition of re-identification. Access will be limited to qualified researchers affiliated with recognized academic or clinical institutions.

DOCUMENTS (1):
  • Study Protocol (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT07311486/Prot_000.pdf